CLINICAL TRIAL: NCT01303120
Title: Does a Single Shot Femoral Nerve Block Alone Produce Appropriate Pain Relief After Total Knee Arthroplasty or Should an Addition of Sciatic, Obturator and Lateral Femoral Cutaneous Nerve Blocks be Recommended?
Brief Title: Does a Single Shot Femoral Nerve Block Alone Produce Appropriate Pain Relief?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: A Stav, MD, Hillel Yaffe Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0021-11-HYMC
Record Dates: First submitted 2011-02-20; First posted 2011-02-24 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2011-02

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Femoral Nerve Block (Active Comparator)
  Interventions: Drug: Femoral Nerve Block
- Combined Nerve Blocks (Active Comparator)
  Interventions: Drug: Combined nerve blocks
- Patient-controlled analgesia (Active Comparator)
  Interventions: Drug: Patient-controlled analgesia

INTERVENTIONS:
Drug: Femoral Nerve Block — Preoperative Bupivacaine 0.5%, perineurally as single shot
  Arms: Femoral Nerve Block
Drug: Combined nerve blocks — Preoperative Bupivacaine 0.5%, perineurally as single shot
  Arms: Combined Nerve Blocks
Drug: Patient-controlled analgesia — Patient controlled analgesia with morphine
  Arms: Patient-controlled analgesia

SUMMARY:
The aim of this study is to compare the efficacy of the analgesic effect of the preoperative femoral nerve block alone versus combined femoral, sciatic, obturator and lateral femoral cutaneous nerve blocks in patients after TKA in the immediate postoperative period.

DETAILED DESCRIPTION:
Bupivacaine will be used for all the nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Undergoing two TKA
* Understanding PCA protocol

Exclusion Criteria:

* Skin infection near injection site
* Allergy to local analgesics
* Peripheral neuropathy
* Coagulopathy
* Dementia
* Proven opioid dependency

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of single short femoral nerve block | Three days

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

REFERENCES:
- [Derived] Stav A, Reytman L, Sevi R, Stav MY, Powell D, Dor Y, Dudkiewicz M, Bayadse F, Sternberg A, Soudry M. Femoral versus Multiple Nerve Blocks for Analgesia after Total Knee Arthroplasty. Rambam Maimonides Med J. 2017 Jan 30;8(1):e0006. doi: 10.5041/RMMJ.10281. PMID 28178436